CLINICAL TRIAL: NCT03119948
Title: Partial Blocks of Rectus Femoris and Soleus With Botulinum Toxin Type A to Improve Gait in Hemiparesis. A Randomized Multicenter Placebo-controlled Trial
Brief Title: Partial Blocks of Rectus Femoris and Soleus With Botulinum Toxin Type A (Xeomin®) to Improve Gait in Hemiparesis
Acronym: GENUFLEX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P101107; 2013-005088-13 (EudraCT Number)
Record Dates: First submitted 2016-12-23; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2016-12

CONDITIONS: Hemiparesis After Stroke; Traumatic Brain Injury
Keywords: Muscle spasticity; Botulinum toxin
MeSH Terms: conditions — Brain Injuries, Traumatic; Muscle Spasticity | interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Placebo Comparator): Placebo in soleus and placebo in rectus femoris, and placebo in additional muscles as per investigator's choice among tibialis posterior, toe flexors (long or short), gastrocnemius muscles or peroneus longus.
  Interventions: Drug: Placebo injection
- Group 2 (Active Comparator): Botulinum toxin type A in soleus and placebo in rectus femoris, and Botulinum toxin type A in additional muscles as per investigator's choice among tibialis posterior, toe flexors (long or short), gastrocnemius muscles or peroneus longus.
  Interventions: Drug: Placebo injection and botulinum toxin injection
- Group 3 (Active Comparator): Botulinum toxin type A in soleus and in rectus femoris, and Botulinum toxin type A in additional muscles as per investigator's choice among tibialis posterior, toe flexors (long or short), gastrocnemius muscles or peroneus longus.
  Interventions: Drug: Botulinum toxin injection

INTERVENTIONS:
Drug: Placebo injection — Placebo in soleus and placebo in rectus femoris, and placebo in additional muscles as per investigator's choice among tibialis posterior, toe flexors (long or short), gastrocnemius muscles or peroneus longus.
  150U (x 7.5 ml) placebo Sol + 150U (x 7.5 ml) placebo RF + 100U (5ml) placebo distributed between tibialis posterior, FHL (flexor hallucis longus), FCB (flexor digitorum brevis), gastrocnemius muscles or peroneus longus, based upon investigator clinical judgment
  Arms: Group 1
Drug: Botulinum toxin injection — Botulinum toxin type A in soleus and in rectus femoris, and Botulinum toxin type A in additional muscles as per investigator's choice among tibialis posterior, toe flexors (long or short), gastrocnemius muscles or peroneus longus.
  150U (x 7.5 ml) Xeomin® 20U/ml Sol + 150U (x 7.5 ml) Xeomin® 20U/ml RF + 100U (5ml) Xeomin® distributed between tibialis posterior, FHL (flexor hallucis longus), FCB (flexor digitorum brevis), gastrocnemius muscles or peroneus longus, based upon investigator clinical judgment.
  Arms: Group 3
Drug: Placebo injection and botulinum toxin injection — Botulinum toxin type A in soleus and placebo in rectus femoris, and Botulinum toxin type A in additional muscles as per investigator's choice among tibialis posterior, toe flexors (long or short), gastrocnemius muscles or peroneus longus..
  150U (x 7.5 ml) Xeomin® 20U/ml Sol + 150U (x 7.5 ml) placebo RF + 100U (5ml) Xeomin® distributed between tibialis posterior, FHL (flexor hallucis longus), FCB (flexor digitorum brevis), gastrocnemius muscles or peroneus longus, based upon investigator clinical judgment.
  Arms: Group 2

SUMMARY:
The most common motor deficiency after stroke or traumatic brain injury is hemiparesis. Most hemiparetic patients recover walking, but rarely with a speed permitting easy ambulation outdoors with family or friends. One of the mechanisms of gait impairment in hemiparesis is insufficient active hip flexion during swing phase, which leads to insufficient ground clearing at swing phase, with associated gait slowness and risks of fall.

The main hypothesis behind the present study is that insufficient hip flexion during hemiparetic gait is partly due to overactivity of rectus femoris. Focal treatment of lower limb muscle overactivity using botulinum toxin has not been demonstrated to increase walking speed in hemiparesis as yet. However, most studies have focused distally, on improving foot dorsiflexion only. The purpose of this study is to compare the effects of botulinum toxin injection and placebo in rectus femoris (RF) + plantar flexors versus plantar flexors only.

DETAILED DESCRIPTION:
Randomized, double blind, parallel-group study in chronic, non-evolutive brain damaged patients (>6 months since stroke or brain trauma) and ambulating at <1.3 m/sec at maximal speed barefoot (AT10) Group 1: 150U (x 7.5 ml) placebo Sol + 150U (x 7.5 ml) placebo RF + 100U (5ml) placebo distributed between tibialis posterior, FHL (flexor hallucis longus), FCB (flexor digitorum brevis), gastrocnemius muscles or peroneus longus, based upon investigator clinical judgment.

Group 2: 150U (x 7.5 ml) Xeomin® 20U/ml Sol + 150U (x 7.5 ml) placebo RF + 100U (5ml) Xeomin® distributed between tibialis posterior, FHL (flexor hallucis longus), FCB (flexor digitorum brevis), gastrocnemius muscles or peroneus longus, based upon investigator clinical judgment.

Group 3: 150U (x 7.5 ml) Xeomin® 20U/ml Sol + 150U (x 7.5 ml) Xeomin® 20U/ml RF + 100U (5ml) Xeomin® distributed between tibialis posterior, FHL (flexor hallucis longus), FCB (flexor digitorum brevis), gastrocnemius muscles or peroneus longus, based upon investigator clinical judgment.

ELIGIBILITY:
Inclusion Criteria

* Hemiparesis from stroke, brain trauma, or non evolutive brain tumor >6 months before enrolment
* Hip flexion at swing phase on the paretic side clinically insufficient (rated <15° by the clinical investigator)
* Passive ankle dorsiflexion clinically insufficient at late stance (rated <90° by the clinical investigator)
* Maximal ambulation speed barefoot over 10 metres < 1,3 m/sec
* Age ≥ 18
* Signed consent form

Exclusion Criteria

* Ambulation impossible barefoot
* Passive hip flexion amplitude (with the knee flexed) < 45° on paretic side
* Severe intercurrent disease ou cognitive dysfunction making effective communication or study participation impossible.
* Current anticoagulation with INR> 3,5 ; less than 15 days prior to D1
* Pregnancy, lactation, or premenopause woman not taking contraception
* Hypersensitivity to botulinum toxin or its excipients, myasthenia gravis, Lambert-Eaton syndrome, concomitant aminoside treatment.
* Infection or inflammation at injection sites.
* Injection in lower limb less than 3 months prior to D1
* Person not covered by social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in maximum speed of barefoot ambulation without technical assistance over 10 meters, between the pre-injection visit (D1) and 3 weeks (D21) post injection | Preinjection visit (D1) and 3 weeks post injection (D21)

SECONDARY OUTCOMES:
Change ambulation speed at comfortable and maximal speed, barefoot and with shoes over 10 meters | Day 1 and Day 21
Maximal amplitude and speed of active hip flexion and passive knee flexion during swing phase, measured in gait kinematic recording, at comfortable and maximal speed | Day 1 and Day 21
Maximal amplitude and speed of passive ankle dorsiflexion at late stance phase, measured in gait kinematic recording, at comfortable and maximal speed | Day 1 and Day 21
Maximal voluntary isometric EMG (MVIE) of rectus femoris and soleus, measured by surface EMG, in an isometric position with hip at 15° flexion, knee at 30° flexion, and ankle at 80° of dorsiflexion | Day 1 and Day 21
  calculating the mean rectified voltage over 100 ms around the peak of rectified EMG on each of these muscles
Mean rectified voltage of rectus femoris and soleus during the first half of swing phase (MRVSP), from toe-off to maximal hip flexion, measured by surface EMG (electrodes 2 cm apart) immediately after MVIE measure. | Day 1 and Day 21
Cocontraction indices of rectus femoris and soleus during the first half of swing phase, calculating the ratio MRVSP/MVIE for each of these muscles. | Day 1 and Day 21
Mean rectified voltage of soleus during the first half of stance phase (MRVSP), from heel-on to maximal knee extension, measured by surface EMG (electrodes 2 cm apart) immediately after MVIE measure. | Day 1 and Day 21
Inappropriate Contraction Indices of soleus during the first half of stance phase, calculating the ratio MRVSP / MVIE | Day 1 and Day 21
Spasticity Angle et grade of rectus femoris and soleus (Five Step Assessment) | Day 1, Day 21, Day 60
Weakness Angle of rectus femoris and soleus (Five Step Assessment) | Day 1, Day 21, Day 60
Quality of life measured by EQ5D | Day 1, Day 60
Mean weekly number of steps | Between Day-15 and Day1, Day7 and Day21 and between Day45 and Day60
Potential AEs of injections (pain or discomfort during the injection or post injection, or ecchymoses at insertion site) and potential AEs related to the injected drug (muscle weakening, allergies) | Day 1, Day 21, Day 60
Step length at comfortable and maximal speed, barefoot and with shoes over 10 meters | Day 1 and Day 21
Step cadence at comfortable and maximal speed, barefoot and with shoes over 10 meters | Day 1 and Day 21
Physiological Cost Index (PCI) over a walking test of 2 minutes at maximal speed with shoes | Day 1 and Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel GRACIES, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Derived] Ghedira M, Albertsen IM, Mardale V, Loche CM, Vinti M, Gracies JM, Bayle N, Hutin E. Agonist and antagonist activation at the ankle monitored along the swing phase in hemiparetic gait. Clin Biomech (Bristol). 2021 Oct;89:105459. doi: 10.1016/j.clinbiomech.2021.105459. Epub 2021 Aug 20. PMID 34438333